CLINICAL TRIAL: NCT01468467
Title: A Phase 1 Study of AC220 (ASP2689) as Maintenance Therapy in Subjects With Acute Myeloid Leukemia Who Have Been Treated With an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: A Study of AC220 Given After Transplant in Subjects With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Ambit Biosciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2689-CL-0011
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-11

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AC220; Acute Myeloid Leukemia (AML); Transplantation; Stem Cell Transplantation; Allogeneic Transplantation; FMS-like tyrosine kinase (FLT3); FMS-like tyrosine kinase (FLT3) Inhibitor; Kinase; Kinase Inhibitor; Pharmacokinetics; ASP2689; quizartinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC220 (Experimental)
  Interventions: Drug: AC220

INTERVENTIONS:
Drug: AC220 — Oral Liquid
  Other Names: quizartinib; ASP2689

SUMMARY:
The purpose of this study is to define a safe dose of AC220 when given as maintenance therapy after treatment with an allogeneic stem cell transplant.

DETAILED DESCRIPTION:
This is a two-part, sequential group dose escalation study.

In Part 1, subjects will be enrolled into successive cohorts to determine the maximum tolerated dose (MTD). Dose escalation decision will be made based on dose limiting toxicities (DLTs) that occur in subjects treated to date at a given dose level. In Part 2, a confirmation cohort will be opened to confirm the safety at the MTD.

Subjects who have had an allogeneic Hematopoietic Stem Cell Transplant (HSCT) will enter treatment with AC220 between 30 to 60 days after receiving allogeneic HSCT. AC220 will be administered every day, with 28 consecutive days defined as a treatment cycle. Subjects may receive up to 24 continuous treatment cycles. Subjects will have study visits each week for the first 2 cycles, and then on Day 1 of each cycle after that.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of acute myeloid leukemia (AML) according to WHO classification (2008) and has received a high dose or a reduced intensity conditioning allogeneic Hematopoietic Stem Cell Transplant (HSCT) during first or second remission and within 30 to 60 days prior to first dose of AC220. Donors may be human leukocyte antigen (HLA)-matched for HLA-A, B, C, DRB1, and DQB1 by high resolution typing, related or unrelated (only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing) Note: more than one HSCT is allowed
* Subject must be in morphologic remission (< 5% marrow blasts) and without active central nervous system (CNS) AML within 14 days prior to first dose of AC220
* Subject must have CD3 donor chimerism > 50 % at Screening
* Subject has a Karnofsky Performance Status (KPS) of ≥ 60
* Subject must have absolute neutrophil count (ANC) > 1000/mm3 and platelet count > 50,000/mm3 without platelet transfusion support within 2 weeks prior to first dose
* Subject must have adequate renal, hepatic, and coagulation parameters
* Female subjects must not be lactating and must not be breastfeeding at Screening or during the study period and for 28 days [or five half lives of the study drug whichever is longer] after final study drug administration.
* Subject is able to comply with study procedures and follow-up examinations

Exclusion Criteria:

* Subject received AC220 and relapsed during treatment with AC220
* Subject has active ≥ Grade 2 graft versus host disease (GVHD)
* Subject has received concurrent chemotherapy, immunotherapy, or radio-therapy within 21 days prior to the first dose of AC220, or any antineoplastic therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation) within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
* Subject requires treatment with concomitant drugs that prolong QT/QTc interval or strong cytochrome P-3A4 (CYP3A4) inhibitors or inducers with the exception of immunosuppressants, antibiotics, antifungals, and antivirals that are used as standard of care post-transplant or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject
* Subject requires treatment with anticoagulant therapy
* Subject has a known positive test for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen
* Subject had major surgery within 4 weeks prior to first dose of AC220
* Subject has uncontrolled or significant cardiovascular disease
* Subject has an active acute fungal, bacterial, or other infection that is unresponsive to therapy
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives whichever is longer, prior to the initiation of Screening.
* Subject has any medical, psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | up to Day 56
  From first dose through last dose of Cycle 2
Safety assessed by recording adverse events, physical examinations, vital signs, electrocardiograms (ECGs) and laboratory assessments | 30 days after last subject discontinues treatment (maximum of 24 months)

SECONDARY OUTCOMES:
Duration of confirmed complete remission (CR) | 24 months
  Time from first dose until date of relapse
Duration of overall complete remission | 24 months
  Complete remission (CR) + CR with incomplete platelet recovery (CRp) + CR with incomplete hematologic recovery (CRi) + complete molecular remission (CRm)
Disease-free survival | 30 days after last subject discontinues treatment (maximum of 24 months)
  Time from first dose until date of relapse or death
Overall survival | 30 days after last subject discontinues treatment (maximum of 24 months)
  Time from first dose until date of death from any cause
Percentage of transplant rejections | 30 days after last subject discontinues treatment (maximum of 24 months)
  Through End of Treatment
Percentage of Subjects with Graft-versus-Host Disease (GVHD) | Up through 24 months of treatment
Percentage of Donor Chimerism | Up through 24 months of treatment
Treatment-related mortality (TRM) | Up through 24 months of treatment
  Death in CR (CR, CRm, CRp and CRi)
Composite of pharmacokinetics: AUC24 , Cmax, Ctrough and Tmax | Up through 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guy Gammon, MB, BS, MRCP, Study Director — Medical Monitor, Ambit Biosciences Corporation
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Northwestern University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - M.D. Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/